CLINICAL TRIAL: NCT02181491
Title: PET Imaging in Cocaine Self Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0811004457
Record Dates: First submitted 2014-07-01; First posted 2014-07-04 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P943 PET Scan (Experimental)
  Interventions: Other: [11C]-P943

INTERVENTIONS:
Other: [11C]-P943

SUMMARY:
There has been recent interest in the role of the 5-HT1B receptor as a possible modulating factor in cocaine dependence, certainly in preclinical models. The Yale Positron Emission Tomography (PET) Center has developed a novel 5-HT1B receptor antagonist radioligand, [11C]-P943, which has been validated in human studies. We hypothesize that the 5-HT1B receptor plays a key role in cocaine dependence. The long term goal of this project would be to study pharmacological manipulation of the 5-HT1B receptor as a potential molecular target for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 50 years
2. voluntary, written, informed consent
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations
4. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (B-HCG) test
5. English speaking
6. No other major Axis DSM-IV diagnosis present, besides required as below

Inclusion criteria for cocaine dependent:

1. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
2. recent street cocaine use
3. intravenous and/or smoked (crack/ freebase) use
4. positive urine toxicology screen for cocaine

Inclusion criteria for healthy controls:

1. No current, or history of, any DSM-IV diagnosis
2. No first-degree relative with history of psychotic, mood, or anxiety disorder

Exclusion Criteria:

1. medical contraindications to AMPT administration (e.g., known sensitivity/reaction to AMPT)
2. medical contraindications to MPH administration (e.g., history of cardiac problems, seizures, etc.)
3. drug or alcohol dependence (except nicotine)
4. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine or pathological gambling
5. positive answers on the cardiac screening questionnaire that may place the subject at higher risk, as determined by cardiologist review of both the questionnaire responses and screening ECG
6. current use of psychotropic and/or potentially psychoactive prescription medication
7. physical or laboratory (B-HCG) evidence of pregnancy
8. clotting disorders or recent anticoagulant therapy
9. MRI-incompatible implants and other contraindications for MRI (i.e., aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker)
10. history of claustrophobia or feeling of inability to lie still on his back for the PET or MRI scans
11. history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over Radioactive Drug Research Committee (RDRC) limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year
12. donation or loss of 550 mL of blood or more (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to the first dose of study drug
13. use any prescription medications and/or over-the-counter medications, vitamins and/or herbal supplements within 2 weeks prior to study and for the duration of the study without approval from the study doctor
14. eat grapefruit or grapefruit products, and drink alcohol, and anything containing caffeine 3 days before study and during study
15. For CD subjects, < 1 year of cocaine dependence
16. Subjects with current, past, or anticipated exposure to radiation in the workplace

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
BPND | 1 week
  BPND is a measure of serotonin receptor availability

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, PhD, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States